CLINICAL TRIAL: NCT04017312
Title: Evaluation of HFCWO Using The Vest® System for Treatment of Non-Cystic Fibrosis Bronchiectasis in the Home Setting
Brief Title: A Pilot Study to Evaluate the Use of the Vest® System for Treatment of Bronchiectasis Patients in the Home Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR-2019-001
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Bronchiectasis; Bronchiectasis With Acute Exacerbation
Keywords: HFCWO; Airway Clearance therapy; PEP; The Vest®; Non Cystic Fibrosis Bronchiectasis; HFCWC; High frequency chest wall oscillation
MeSH Terms: conditions — Bronchiectasis | interventions — Chest Wall Oscillation

STUDY DESIGN:
Intervention Model Description: The study will be a non-blinded prospective Randomized Control Trial (RCT) pilot study with subjects requiring airway clearance therapy randomized to Oscillating Positive Expiratory Pressure (OPEP) therapy as the control group and High Frequency Chest Wall Oscillation (HFCWO) therapy as the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HFCWO group (Active Comparator): Subjects in this arm of treatment will use The Vest® as their primary airway clearance modality for the duration of the study.
  Interventions: Device: High Frequency Chest Wall Oscillation
- OPEP group (Active Comparator): Subjects in this arm of treatment will use the Acapella® as their primary airway clearance modality for the duration of the study.
  Interventions: Device: Oscillating Positive Expiratory Pressure (OPEP)

INTERVENTIONS:
Device: High Frequency Chest Wall Oscillation — High frequency chest wall oscillation (HFCWO) therapy (also known as high-frequency chest-wall compression or HFCWC) is commonly prescribed to provide routine airway clearance in patients with bronchiectasis as well as other patients with a need for regular airway clearance therapy. HFCWO generates high velocity expiratory airflow. This airflow is thought to mobilize secretions by the sheer force created, effecting changes in rheology and moving mucus in a cephalad direction during the oscillation. The Vest® Airway Clearance System, a commonly used device, generates HFCWO using an air pulse generator and an inflatable garment that delivers pressure pulses to the thorax. These pressure pulses within the garment create HFCWO.
  Other Names: The Vest® Airway Clearance System
  Arms: HFCWO group
Device: Oscillating Positive Expiratory Pressure (OPEP) — Oscillating PEP is an airway clearance technique, where the person blows all the way out many times through a device. These types of oscillating PEP devices work in two ways. Firstly, they use resistance to make it more difficult during the breath out, like non-oscillating PEP devices. Oscillating PEP devices also create vibrations when breathing out. The vibrations move mucus from the surface of the airways. After blowing through the device several times, the person will huff and cough to clear the mucus from the lungs.
  Other Names: Acapella®
  Arms: OPEP group

SUMMARY:
This a 70 patient multi-site non blinded randomized control trial evaluating the use of the Vest® System for treatment of Non-Cystic Fibrosis Bronchiectasis (NCFBE) patients in the home setting. The study will assess outcomes in subjects requiring airway clearance therapy randomized to Oscillating Positive Expiratory Pressure (OPEP) therapy as the control group and High Frequency Chest Wall Oscillation (HFCWO) therapy as the intervention group

DETAILED DESCRIPTION:
Patients with NCFBE who require regular home airway clearance therapy will be eligible to be screened for inclusion in the study.

After enrollment, baseline data including demographics, pulmonary related medical history including acute exacerbations (pulmonary-related hospitalizations, ED visits and physician office visits) will be collected Pulmonary function tests (PFTs) (spirometry), and a six-minute walk test will be completed. Quality of Life measures and inflammatory markers and will be collected.

Patients will be randomized to HFCWO or OPEP therapy. Each device will be used within the approved product labeling. These will be the primary airway clearance devices for these patients during the 12 months of the study period.

Following enrollment in the study and completion of a baseline visit, subjects will be seen for follow-up visits.

Detailed documentation of health status and medical history will be collected during the 12-month study period and/or at each study visit to document the occurrence of acute exacerbations and to determine time to first exacerbation, number of hospitalizations and hospitalization days, number of ICU admissions and ICU days, and number of outpatient visits (Physician's office visit, Urgent Care Visits, ED visits)

At 3 months, 6 months and 12 months following the baseline visit, the following tests/procedures will be performed. At each follow-up study visit:

* Acute exacerbations that occurred during the prior 3-month period will be documented/verified
* Pulmonary function will be assessed using standard spirometry to obtain FEV1, FVC and FEV1/FVC.
* 6-minute walk test will be completed to assess respiratory status and endurance
* The QoL-B quality of life survey will be conducted
* A sputum sample will be collected. Sputum samples will be transported to a central lab to test for inflammatory markers (sputum neutrophil elastase in μg/ml).

Mean adherence to the prescribed treatment regimen will be collected and assessed using the validated Modified Self-Reported Medication-Taking Scale. Adherence data in the HFCWO arm will also be collected via the VisiView patient portal.

Adherence results will be collected at the 3-month visit, 6-month visit and 12-month visits.

Any device related adverse events which occur after initial therapy with The Vest® System or Acapella therapy will be recorded.

Any equipment related complaints which occur after initial therapy with The Vest® System or Acapella therapy will be recorded.

At the end of the 12-month study period, all subjects will be given the option of receiving HFCWO therapy for additional 6 month follow up period with outcomes data assessed at the 15-month and 18-month (from baseline visit) time points.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of Bronchiectasis based on high resolution chest CT scan
* History of at least 2 acute exacerbations or hospitalizations in the past 12 months
* Clinically stable for >2 weeks prior to study entry
* FEV1 >30% predicted
* Age18-80 years
* Signed informed consent

Exclusion Criteria:

* Diagnosis of Cystic Fibrosis
* History of bronchiectasis secondary to primary immunodeficiency
* Active pulmonary tuberculosis
* Active treatment of Non-Tuberculous Mycobacterium (NTM)
* Patients currently on home HFCWO treatment or home HFCWO treatment within the past 24 months
* Diagnosed comorbidity or medical indication that would prevent study completion
* History of pneumothorax within past 6 months
* History of hemoptysis requiring embolization within past 12 months
* Inability to perform HFCWO therapy or OPEP therapy as directed
* Pregnancy or lactation
* Inability or unwillingness to complete study visits or provide follow-up data as required by the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Frequency of acute exacerbations of bronchiectasis | 12 months
  Acute exacerbation periods will be defined as per the European Respiratory Society consensus definition:
  * A deterioration in three or more of the following key symptoms for at least 48 h:
    * Cough
    * Sputum volume and/or consistency
    * Sputum purulence
    * Breathlessness and/or exercise tolerance
    * Fatigue and/or malaise;
    * Hemoptysis AND
  * A clinician determines that a change in bronchiectasis treatment is required

SECONDARY OUTCOMES:
6-minute walk test | 12 months
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise. It will provide information regarding functional capacity and response to therapy.
Pulmonary function tests | 12 months
  FVC, FEV1 and FEV1/FVC as indicators of pulmonary function will be assessed using standard spirometry
Quality of life measure using the Quality of Life - Bronchiectasis (QoL-B) tool | 12 months
  The Quality of Life-Bronchiectasis (QoL-B), a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with NCFBE, contains 37 items on 8 scales (Respiratory Symptoms, Physical, Role, Emotional and Social Functioning, Vitality, Health Perceptions and Treatment Burden)
Time to first exacerbation | 12 months
  The duration of time from initiation of therapy to occurrence of an episode of acute exacerbation of bronchiectasis
Number of exacerbation related hospitalizations | 12 months
  This is the total number of times the subject was admitted as an inpatient due to symptoms of an acute exacerbation
Number of exacerbation related inpatient hospital days | 12 months
  This is the total number of days the subject spent in an inpatient non-ICU setting due to symptoms of an acute exacerbation
Number of exacerbation related ICU admissions | 12 months
  This is the total number of times the subject got admitted into an ICU facility due to symptoms of an acute exacerbation
Number of exacerbation related ICU days | 12 months
  This is the total number of days the subject spent in an ICU due to symptoms of an acute exacerbation
Number of exacerbation related outpatient visits (Physician's office, Urgent Care Visits, ED visits) | 12 months
  This is the total number of times the subject visited an outpatient healthcare facility due to symptoms of an acute exacerbation
Number of courses of antibiotics during episodes of acute exacerbation | 12 months
  This is the total courses of antibiotics prescribed for acute exacerbations
Number of antibiotic use days during episodes of acute exacerbation | 12 months
  This is the total number of days spent on antibiotics for acute exacerbations
Mean adherence to prescribed treatment regimen | 12 months
  Adherence data will be collected using the Modified Self-Reported Medication Taking Scale and verified via the VisiView patient portal
Bronchiectasis related medication | 12 months
  Bronchiectasis related medication data will be collected from subject's electronic medical chart

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Basavaraj, MD, Principal Investigator — New York University Langone Health; Clyde Southwell, MD, Principal Investigator — Tennessee Comprehensive Lung and Sleep Center; Julie Philley, MD, Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - Tennessee Comprehensive Lung and Sleep Center, Nashville, Tennessee
  - UT Tyler Health Science Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No